CLINICAL TRIAL: NCT06728813
Title: Assessing the Link Between the Eat-Lancet Index and Sustainable Eating Practices Across Occupational Groups
Brief Title: Eat-Lancet Index and Sustainable Eating Across Professions
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Emine Elibol, Assist. Prof., Ankara Yildirim Beyazıt University
Other Study IDs: AYBUELİBOL006
Record Dates: First submitted 2024-12-03; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Working Adults
Keywords: Sustainability; occupation; healthy eating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Working adults: The study included 2,705 individuals aged 19-65 working in various occupations. Data were collected using a demographic structure survey and the Behaviors Scale Towards Sustainable Nutrition (BSSN). A food consumption frequency survey was administered to calculate the EAT-Lancet Index. Occupations were classified into five groups according to the International Standard Classification of Occupations (ISCO)-88: Groups 1-2, 3-4, 5-8, 6-7, and 9-10. Additionally, occupational skill levels were categorized into four levels (1 being the lowest and 4 the highest) based on ISCO-88.

SUMMARY:
This study aims to evaluate the relationship between the EAT-Lancet Index of occupational groups and sustainable nutrition behaviors. The study included 2,705 individuals aged 19-65 working in various occupations, using dietary assessment tools and the ehaviors Scale Towards Sustainable Nutrition (BSSN), and were analyzed with SPSS 24.

DETAILED DESCRIPTION:
The study included 2,705 individuals aged 19-65 working in various occupations. Data were collected using a demographic structure survey and the Behaviors Scale Towards Sustainable Nutrition (BSSN). A food consumption frequency survey was administered to calculate the EAT-Lancet Index. Occupations were classified into five groups according to the International Standard Classification of Occupations (ISCO)-88: Groups 1-2, 3-4, 5-8, 6-7, and 9-10. Additionally, occupational skill levels were categorized into four levels (1 being the lowest and 4 the highest) based on ISCO-88. Statistical analysis was performed using SPSS version 24.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 to 65 years

Exclusion Criteria:

* Unemployed and retired individuals
* Individuals with alcohol or drug addiction
* Individuals diagnosed with psychiatric or neurological diseases
* Illiterate individuals.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample in Türkiye
Sampling Method: Non-Probability Sample
Enrollment: 2705 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
EAT-Lancet Index score | Baseline
  Food components in the EAT-Lancet diet are classified as "restricted foods" and "emphasized foods." Restricted foods include pork, beef, lamb, poultry, potatoes, eggs, and added sugar. Emphasized foods include fruits, vegetables, legumes, unsaturated fats, fish, whole grains, and nuts. Dietary intake is assessed based on the reported amounts in grams per day of uncooked weight, aligning with the target intake levels specified in the EAT-Lancet diet.
  The index consists of 14 food components, with each scored from 0 to 3. A score of 0 indicates low adherence to the target for a given food component, while a score of 3 reflects high adherence. The total index score ranges from 0 (no adherence) to 42 (perfect adherence, calculated as 14 components × 3 points). The food consumption frequency method was used to calculate the EAT-Lancet Index.

SECONDARY OUTCOMES:
Behaviors scale towards sustainable nutrition (BSSN) score | Baseline
  The scale was developed to measure sustainable consumption behaviors. It consists of 11 questions in total and uses a 7-point Likert format. The scale is divided into two subsections that assess individuals' nutrition and purchasing preferences. A minimum of 0 and a maximum of 66 points are obtained from the scale. Higher scores on the scale indicate stronger sustainable food consumption behaviors.
Sociodemographic characteristics | Baseline
  Sociodemographic characteristics will be assessed using a structured questionnaire developed by the researchers. The questionnaire will include items measuring age, gender, education level, and income status. The results will be presented as numbers and percentages for each characteristic.
Body Mass Index (BMI) | Baseline
  Kilograms per square meter (kg/m2)
Body weight | Baseline
  Body weight in kg
Height | Baseline
  Height in cm

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No